CLINICAL TRIAL: NCT05476848
Title: Evaluation of Oral Health Status and Cytokine Levels in Sars-Cov-2 Hospitalized Patients: A Randomized Clinical Trial
Brief Title: Relationship Between Oral Findings and Salivary Factors in Sars-Cov-2 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Dokuz Eylul University (Other); Izmir Katip Celebi University (Other); Gazi University (Other); Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Cem Peskersoy, Assisstant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 21-6.1T/70
Record Dates: First submitted 2022-05-25; First posted 2022-07-27 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Decay, Dental; Missing Teeth; COVID-19; Cytokine Storm
MeSH Terms: conditions — Dental Caries; Anodontia; COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Care provider, investigator and outcome assessors are chosen from separate specialists (Intensive Care Unit, Dentistry, Infectious Disease Departments).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covid-19 (+) Patients (Experimental): Oral Examination, Radiography, oral (salivary) swap sample collection will be performed.
  Interventions: Diagnostic Test: ELISA test for Cytokines
- Healthy Individuals (Active Comparator): Oral Examination, Radiography, oral (salivary) swap sample collection will be performed.
  Interventions: Diagnostic Test: ELISA test for Cytokines

INTERVENTIONS:
Diagnostic Test: ELISA test for Cytokines — ELISA tests specific for cytokines (IL-1, IL-6, IL-10) and immunoglobulins (IgA, IgG, IgM) will be performed by a biochemistry lab, both for blood samples and oral swap samples.

SUMMARY:
Two hundred individuals will be formed according to the study and control groups: Group-1: coronavirus 2 (Covid-19) (+) patients (n=100) and Group-2: Healthy individuals (in which the volunteers will be included due to group-1) (n=100). Oral examinations including DMFT scores, salivary flow rate, visible gingival index scores and radiographs (OPG) will be performed on both groups on the 1st appointment. Oral swap samples will be collected with sterile swap brushes (Six sample for each person) on the 1st, 7th and 30th days to evaluate the salivary immunoglobulins (Immunoglobulin A (IgA), Immunoglobulin G (IgG), Immunoglobulin M (IgM)) and cytokine (IL-1, IL-6, IL-10) levels. Blood samples will be collected to validate the oral swap test results.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2) is the virus responsible for coronavirus disease 2019 (COVID-19) which also affects all systems of the body including the oral environment. Recent studies have demonstrated the association between oral health status and systemic diseases. including systemic infections and respiratory diseases. Aim of this study is to analyze the immunoglobulin and cytokine levels of SARS-CoV-2 patients and correlate the oral health status of these patients. Our hypotheses are, 1) Covid-19 affects individuals with low oral hygiene (high DMFT score) more severely, 2) Oral cytokine levels will increase similarly to blood levels in patients with Covid-19, 3) Oral immunoglobulin levels in patients with Covid-19 decreased similarly to those in blood. Oral examination of 100 Covid (+) patients which were hospitalized due to acute respiratory failure will be performed in the dental department of each faculty hospital. Decay-Missing-Filled Tooth (DMFT) scores, visible gingival plaque index (Löe-Silness), Bleeding on Probing (BoP) scores, and orthopantomographs (OPG) will be collected for each participant. Oral swap specimens will be collected (6 sample for each person) to evaluate the levels of salivary immunoglobulins (IgA, IgG, IgM) and cytokines (IL-1, IL-6, IL-10) on 1st, 7th, and 30th days. ELISA test will be performed for immunological analysis with ready-made kits (SunRed Biotech. Co, Shanghai, China). Full blood analyses will be performed to validate and correlate the actual cytokine and immunoglobulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Covid (+) patients,
* Patients who were hospitalized due to Acute Respiratory Deficiency,
* Conscious patients in ICU (intensive care unit) or IDMC (Infectious Diseases and Microbiology Clinic).

Exclusion Criteria:

* Patients with Cancer,
* Patients with Autoimmune System diseases,
* Pregnant women,
* Patients with Immune Deficiency diseases (Acquired immune deficiency syndrome - AIDS, Autoimmune lymphoproliferative syndrome - ALPS , Chronic granulomatous disease - CGD, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
DMF Index | Baseline (1st appointment)
  Decay, Missing, Filled teeth scores will be recorded and evaluated for both study groups.
Dental Plaque Status - GI | Baseline (1st appointment), 7th day (2nd appointment), 30th day (3rd appointment)
  Gingival Index scores (visible dental plaque) will be evaluated for both study groups.
Periodontal Bleeding Status - BoP | Baseline (1st appointment), 7th day (2nd appointment), 30th day (3rd appointment)
  Bleeding volume (ml/sec) on probing will be evaluated for both study groups.
Salivary Flow Rate | Baseline (1st appointment), 7th day (2nd appointment), 30th day (3rd appointment)
  Salivary flow rate of each participant is calculated by measuring the unstimulated saliva volume (ml/min).
Oral Cytokine Levels | Baseline (1st appointment), 7th day (2nd appointment), 30th day (3rd appointment)
  Oral cytokine levels will be evaluated for both study groups three times, due to the half-life of specific markers (IL-1, IL-6, IL-10).
Oral Immunoglobulin Levels | Baseline (1st appointment), 7th day (2nd appointment), 30th day (3rd appointment)
  and immunoglobulin levels will be evaluated for both study groups three times, due to the half-life of specific markers (IgA, IgG, IgM).

SECONDARY OUTCOMES:
Age Range of the Participants | Baseline (1st appointment)
  The age distributions of the participants in the study will be recorded, so that it will be examined which age group is affected the most from Covid-19 disease (min age: 18, max age 80).
Gender Distribution | Baseline (1st appointment)
  The gender distributions of the participants in the study will be recorded, so that it will be examined which gender group is affected the most from Covid-19 disease.
Systemical Diseases | Baseline (1st appointment)
  The systemic diseases of the participants in the study will be recorded so that it will be examined with which systemic disease the Covid-19 disease can be most associated.

CONTACTS AND LOCATIONS:
Overall Officials: Cem Peskersoy, Principal Investigator — Ege University Faculty of Dentistry
Locations (4):
- Turkey (Türkiye) (4):
  - Gazi University, Ankara
  - Ege University, Izmir
  - Izmir Katip Celebi University, Izmir
  - Dokuz Eylul University, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peskersoy C, Oguzhan A, Gurlek O. The Effect of Flowable Composite Resins on Periodontal Health, Cytokine Levels, and Immunoglobulins. Biomed Res Int. 2022 Apr 23;2022:6476597. doi: 10.1155/2022/6476597. eCollection 2022. PMID 35502340
- [Background] Peskersoy C, Peker S, Kaya A, Unalp A, Gokay N. Evaluation of the relationship between migraine disorder andoral comorbidities: multicenter randomized clinical trial. Turk J Med Sci. 2016 Apr 19;46(3):712-8. doi: 10.3906/sag-1412-71. PMID 27513246
- [Background] Alfaifi A, Sultan AS, Montelongo-Jauregui D, Meiller TF, Jabra-Rizk MA. Long-Term Post-COVID-19 Associated Oral Inflammatory Sequelae. Front Cell Infect Microbiol. 2022 Mar 2;12:831744. doi: 10.3389/fcimb.2022.831744. eCollection 2022. PMID 35310855